CLINICAL TRIAL: NCT00432380
Title: Immunogenicity and Safety of Two Doses of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Liquid Vaccine (GSK 357941A) in Healthy Infants.
Brief Title: A Study to Evaluate Immune Response and Safety of Two Doses of GSK Biologicals' HRV Liquid Vaccine in Healthy Infants.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109216; 2015-001544-11 (EudraCT Number)
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Infections, Rotavirus; Rotavirus Vaccines
Keywords: Placebo; Double blind; Gastroenteritis; Randomized; Oral live attenuated human rotavirus liquid vaccine
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- PLACEBO-ROTARIX-ROTARIX GROUP (Experimental): Healthy male or female infants between, and including, 5 to 10 weeks of age, were administered 2 oral doses of Rotarix™ liquid vaccine at Month 1 and Month 2, and a single oral dose of placebo at Day 0. Subjects also received routine infant vaccinations according to the Expanded Program of Immunization (EPI) recommendations in Philippines.
  Interventions: Biological: Rotarix™; Biological: Placebo
- ROTARIX-PLACEBO-ROTARIX GROUP (Experimental): Healthy male or female infants between, and including, 5 to 10 weeks of age, were administered 2 oral doses of Rotarix™ liquid vaccine at Day 0 and Month 2, and a single oral dose of placebo at Month 1. Subjects also received routine infant vaccinations according to the Expanded Program of Immunization (EPI) recommendations in Philippines.
  Interventions: Biological: Rotarix™; Biological: Placebo
- PLACEBO GROUP (Placebo Comparator): Healthy male or female infants between, and including, 5 to 10 weeks of age, were administered 3 oral doses of placebo at Day 0, Month 1 and Month 2. Subjects also received routine infant vaccinations according to the Expanded Program of Immunization (EPI) recommendations in Philippines.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix™ — oral doses
  Arms: PLACEBO-ROTARIX-ROTARIX GROUP; ROTARIX-PLACEBO-ROTARIX GROUP
Biological: Placebo — oral dose

SUMMARY:
This study will provide data on the immune response and safety of GSK Biologicals' HRV liquid vaccine when given along with the routine infant immunizations in Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants between, and including, 5-10 weeks of age at the time of the first dose of HRV liquid vaccine or placebo.
* Birth weight of the subject should be > 2000 grams.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol except for DTPw, HBV and OPV vaccines within 14 days before each dose of HRV liquid vaccine or placebo and ending 14 days after. BCG is administered at birth according to the local EPI.
* Concurrently participating in another clinical study, at any time during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the HRV liquid vaccine or placebo.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 5 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2007-03-09 (Actual); Primary Completion 2007-09-04 (Actual); Study Completion 2007-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=273

REFERENCES:
- [Background] Anh DD, Carlos CC, Thiem DV, Hutagalung Y, Gatchalian S, Bock HL, Smolenov I, Suryakiran PV, Han HH. Immunogenicity, reactogenicity and safety of the human rotavirus vaccine RIX4414 (Rotarix) oral suspension (liquid formulation) when co-administered with expanded program on immunization (EPI) vaccines in Vietnam and the Philippines in 2006-2007. Vaccine. 2011 Mar 3;29(11):2029-36. doi: 10.1016/j.vaccine.2011.01.018. Epub 2011 Jan 21. PMID 21256876
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109216 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Period: Overall Study
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Started | 150 | 150 | 75
Completed | 146 | 146 | 74
Not Completed | 4 | 4 | 1
Not completed — Migrated/moved from study area | 3 | 4 | 1
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 150 | 150 | 75 | 375
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.6 (1.07) | 6.5 (1) | 6.6 (1.02) | 6.56 (1.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 76 | 40 | 175
  Male | 91 | 74 | 35 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-rotavirus (Anti-RV) Immunoglobulin A (IgA) Antibody
Description: Seroconversion was defined as the appearance of anti-RV IgA antibody concentrations greater than or equal to (≥) 20 units per milliliter (U/mL) in subjects initially (i.e. prior to the first dose of Rotarix™ vaccine or placebo) seronegative, when administered concomitantly with the second and third routine EPI immunization. This outcome measure only concerns subjects in the Placebo-Rotarix-Rotarix Group.
Time Frame: At Month 3
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all subjects who were seronegative for anti-RV IgA antibodies on the day of Dose 1 of Rotarix™ liquid vaccine or placebo and for whom immunogenicity data were available, at pre-sampling and post-sampling time points.
Measure: Number; unit: Subjects
Arm/Group | Placebo-Rotarix-Rotarix Group
Number analyzed (Participants) | 120
Subjects | 84

2. Secondary Outcome: Number of Seroconverted Subjects for Anti-RV IgA Antibody
Description: Seroconversion was defined as the appearance of anti-RV IgA antibody concentrations ≥ 20 U/mL in subjects initially (i.e. prior to the first dose of Rotarix™ vaccine or placebo) seronegative, when administered concomitantly with the first and third routine EPI immunization. This outcome measure only concerns subjects in the Rotarix-Placebo-Rotarix Group.
Time Frame: At Month 3
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all subjects who were seronegative for anti-RV IgA antibodies on the day of Dose 1 of Rotarix™ liquid vaccine or placebo and for whom immunogenicity data were available, at pre-sampling and post-sampling time points.
Measure: Number; unit: Subjects
Arm/Group | Rotarix-Placebo-Rotarix Group
Number analyzed (Participants) | 120
Subjects | 71

3. Secondary Outcome: Serum IgA Antibody Concentrations Against Rotavirus
Description: Antibody concentrations were presented as geometric mean concentrations (GMCs), expressed in units per milliliter (U/mL). This outcome measure only concerns subjects in Placebo-Rotarix-Rotarix and Rotarix-Placebo-Rotarix Groups.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group
Number analyzed (Participants) | 120 | 120
U/mL | 68 [50.1 to 92.1] | 75.6 [52.5 to 109]

4. Secondary Outcome: Number of Subjects Reporting Grade 2 or Grade 3 Fever, Vomiting or Diarrhea
Description: Any symptom = occurrence of the symptom (i.e. fever or vomiting or diarrhea) regardless of intensity grade or relationship to vaccination. Grade 2 fever = rectal temperature greater than (>) 38.5 - less than or equal to (≤) 39.5degrees Celsius (°C) or axillary temperature > 38.0 - ≤ 39.0°C. Grade 3 fever = rectal temperature > 39.5°C or axillary temperature > 39.0°C. Grade 2 vomiting = 2 episodes of vomiting/ day. Grade 3 vomiting = 3 or more episodes of vomiting/ day. Grade 2 diarrhea = 4-5 looser than normal stools/ day. Grade 3 diarrhea = 6 or more looser than normal stools/ day.
Time Frame: During the 8-day (Days 0-7) period following each dose of study vaccine or placebo and across doses
Population: The analysis was performed on the Total vaccinated Cohort, which included all vaccinated subjects with at least one study vaccine/placebo administration documented.
Measure: Number; unit: Subjects
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Number analyzed (Participants) | 150 | 150 | 75
Subjects
  Any symptom, Dose 1 [N=150, 150, 75] | 57 | 68 | 35
  Any symptom, Dose 2 [N=149, 147, 75] | 52 | 36 | 19
  Any symptom, Dose 3 [N= 146, 147, 75] | 29 | 38 | 24
  Any symptom, Across doses [N= 150, 150, 75] | 86 | 91 | 48

5. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were cough/runny nose, diarrhea, fever (rectally), irritability, loss of appetite and vomiting. Any = any solicited symptom irrespective of intensity grade or relationship to vaccination. Grade 3 cough/runny nose = cough/runny nose which prevented daily activity. Grade 2 diarrhea: 4-5 looser than normal stools/ day. Grade 3 diarrhea = ≥ 6 looser than normal stools/ day. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 2 vomiting= 2 episodes of vomiting/ day. Grade 3 vomiting = ≥ 3 episodes of vomiting/ day. Related = symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: During the 8-day (Days 0-7) period following each dose of study vaccine or placebo and across doses
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Number analyzed (Participants) | 150 | 150 | 75
Subjects
  Any Cough/ runny nose, D1 [N=150, 150, 75] | 52 | 44 | 23
  Grade 3 Cough/ runny nose, D1 [N=150, 150, 75] | 0 | 1 | 1
  Related Cough/ runny nose, D1 [N=150, 150, 75] | 1 | 0 | 1
  Any Diarrhea, D1 [N=150, 150, 75] | 5 | 4 | 6
  Grade 3 Diarrhea, D1 [N=150, 150, 75] | 2 | 0 | 0
  Related Diarrhea, D1 [N=150, 150, 75] | 5 | 4 | 5
  Any Fever, D1 [N=150, 150, 75] | 122 | 117 | 54
  Grade 3 Fever, D1 [N=150, 150, 75] | 3 | 5 | 0
  Related Fever, D1 [N=150, 150, 75] | 121 | 114 | 53
  Any Irritability, D1 [N=150, 150, 75] | 87 | 72 | 34
  Grade 3 Irritability, D1 [N=150, 150, 75] | 3 | 5 | 0
  Related Irritability, D1 [N=150, 150, 75] | 81 | 70 | 34
  Any Loss of appetite, D1 [N=150, 150, 75] | 26 | 35 | 17
  Grade 3 Loss of appetite, D1 [N=150, 150, 75] | 1 | 0 | 0
  Related Loss of appetite, D1 [N=150, 150, 75] | 20 | 31 | 15
  Any Vomiting, D1 [N=150, 150, 75] | 32 | 24 | 5
  Grade 3 Vomiting, D1 [N=150, 150, 75] | 2 | 1 | 2
  Related Vomiting, D1 [N=150, 150, 75] | 23 | 21 | 5
  Any Cough/ runny nose, D2 [N=149, 147, 75] | 48 | 37 | 21
  Grade 3 Cough/ runny nose, D2 [N=149, 147, 75] | 2 | 0 | 1
  Related Cough/ runny nose, D2 [N=149, 147, 75] | 0 | 0 | 1
  Any Diarrhea, D2 [N=149, 147, 75] | 3 | 1 | 0
  Grade 3 Diarrhea, D2 [N=149, 147, 75] | 1 | 0 | 0
  Related Diarrhea, D2 [N=149, 147, 75] | 1 | 1 | 0
  Any Fever, D2 [N=149, 147, 75] | 103 | 94 | 45
  Grade 3 Fever, D2 [N=149, 147, 75] | 3 | 4 | 2
  Related Fever, D2 [N=149, 147, 75] | 102 | 93 | 45
  Any Irritability, D2 [N=149, 147, 75] | 55 | 45 | 24
  Grade 3 Irritability, D2 [N=149, 147, 75] | 0 | 0 | 0
  Related Irritability, D2 [N=149, 147, 75] | 52 | 43 | 24
  Any Loss of appetite, D2 [N=149, 147, 75] | 20 | 21 | 8
  Grade 3 Loss of appetite, D2 [N=149, 147, 75] | 0 | 0 | 1
  Related Loss of appetite, D2 [N=149, 147, 75] | 16 | 20 | 7
  Any Vomiting, D2 [N=149, 147, 75] | 15 | 17 | 5
  Grade 3 Vomiting, D2 [N=149, 147, 75] | 0 | 1 | 0
  Related Vomiting, D2 [N=149, 147, 75] | 11 | 14 | 4
  Any Cough/ runny nose, D3 [N=146, 147, 75] | 36 | 31 | 23
  Grade 3 Cough/ runny nose, D3 [N=146, 147, 75] | 0 | 6 | 1
  Related Cough/ runny nose, D3 [N=146, 147, 75] | 0 | 0 | 0
  Any Diarrhea, D3 [N=146, 147, 75] | 2 | 1 | 1
  Grade 3 Diarrhea, D3 [N=146, 147, 75] | 0 | 0 | 0
  Related Diarrhea, D3 [N=146, 147, 75] | 2 | 1 | 1
  Any Fever, D3 [N=146, 147, 75] | 91 | 91 | 48
  Grade 3 Fever, D3 [N=146, 147, 75] | 3 | 5 | 2
  Related Fever, D3 [N=146, 147, 75] | 87 | 89 | 47
  Any Irritability, D3 [N=146, 147, 75] | 33 | 40 | 21
  Grade 3 Irritability, D3 [N=146, 147, 75] | 0 | 3 | 2
  Related Irritability, D3 [N=146, 147, 75] | 31 | 38 | 20
  Any Loss of appetite, D3 [N=146, 147, 75] | 19 | 18 | 7
  Grade 3 Loss of appetite, D3 [N=146, 147, 75] | 0 | 1 | 0
  Related Loss of appetite, D3 [N=146, 147, 75] | 19 | 17 | 7
  Any Vomiting, D3 [N=146, 147, 75] | 10 | 8 | 1
  Grade 3 Vomiting, D3 [N=146, 147, 75] | 0 | 2 | 0
  Related Vomiting, D3 [N=146, 147, 75] | 8 | 4 | 1
  Any Cough/runny nose, Across [N=150, 150, 75] | 82 | 69 | 40
  Grade 3 Cough/runny nose, Across [N=150, 150, 75] | 2 | 6 | 2
  Related Cough/runny nose, Across [N=150, 150, 75] | 1 | 0 | 2
  Any Diarrhea, Across [N=150, 150, 75] | 8 | 6 | 7
  Grade 3 Diarrhea, Across [N=150, 150, 75] | 3 | 0 | 0
  Related Diarrhea, Across [N=150, 150, 75] | 6 | 6 | 6
  Any Temperature, Across [N=150, 150, 75] | 139 | 137 | 69
  Grade 3 Temperature, Across [N=150, 150, 75] | 8 | 13 | 3
  Related Temperature, Across [N=150, 150, 75] | 138 | 135 | 69
  Any Irritability, Across [N=150, 150, 75] | 93 | 78 | 40
  Grade 3 Irritability, Across [N=150, 150, 75] | 3 | 7 | 2
  Related Irritability, Across [N=150, 150, 75] | 90 | 76 | 40
  Any Loss of appetite, Across [N=150, 150, 75] | 40 | 46 | 23
  Grade 3 Loss of appetite, Across [N=150, 150, 75] | 1 | 1 | 1
  Related Loss of appetite, Across [N=150, 150, 75] | 35 | 42 | 21
  Any Vomiting, Across [N=150, 150, 75] | 35 | 32 | 9
  Grade 3 Vomiting, Across [N=150, 150, 75] | 2 | 3 | 2
  Related Vomiting, Across [N=150, 150, 75] | 27 | 26 | 8

6. Secondary Outcome: Number of Subjects Reporting RV in Gastroenteritis (GE) Episodes
Description: Presence of RV (vaccine strain or wild-type) in GE stools.
Time Frame: From Dose 1 of study vaccine or placebo (at Day 0) up to Month 3
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Number analyzed (Participants) | 150 | 150 | 75
Subjects
  Between Dose 1 and before Dose 2 [N=150, 150, 75] | 1 | 0 | 1
  Between Dose 2 and before Dose 3 [N=149, 147, 75] | 0 | 0 | 0
  Between Dose 3 and Month 3 [N=146, 147, 75] | 0 | 0 | 0
  Between Dose 1 and Month 3 [N=150, 150, 75] | 1 | 0 | 1

7. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Event (AE)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Any solicited symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 31-day (Days 0-30) period following any study vaccine dose or placebo
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Number analyzed (Participants) | 150 | 150 | 75
Subjects | 53 | 60 | 19

8. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include any untoward medical occurrences that results in death, are life threatening, requires hospitalization or prolongation of hospitalization, result in disability/incapacity or congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (from Day 0 to Month 3)
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Number analyzed (Participants) | 150 | 150 | 75
Subjects | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Solicited symptoms were collected during the 8-day (Days 0-7) post-vaccination period. Unsolicited AEs were collected during the 31-day (Days 0-30) post-vaccination period. SAEs were collected throughout the entire study period (Months 0 to 3).
Arm/Group | Placebo-Rotarix-Rotarix Group | Rotarix-Placebo-Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 1/150 | 1/150 | 1/75
Other Adverse Events (participants affected / at risk) | 139/150 | 137/150 | 69/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Rotarix-Rotarix Group (N=150) | Rotarix-Placebo-Rotarix Group (N=150) | Placebo Group (N=75)
Milk allergy (Immune system disorders) | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Rotarix-Rotarix Group (N=150) | Rotarix-Placebo-Rotarix Group (N=150) | Placebo Group (N=75)
Cough/runny nose (General disorders) | 82 | 69 | 40
Diarrhea (General disorders) | 8 | 6 | 7
Fever (Rectally) (General disorders) | 139 | 137 | 69
Irritability (General disorders) | 93 | 78 | 40
Loss of appetite (General disorders) | 40 | 46 | 23
Vomiting (General disorders) | 35 | 32 | 9
Upper respiratory tract infection (Infections and infestations) | 19 | 21 | 6
Rhinitis (Infections and infestations) | 13 | 16 | 6
Bronchitis (Infections and infestations) | 7 | 7 | 4
Diarrhea infectious (Infections and infestations) | 5 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.